CLINICAL TRIAL: NCT04215588
Title: Heparin and Protamine Titration Using Optical Detection Technology in Patients Undergoing Cardiac Surgery Under Minimal Invasive Extracorporeal Circulation
Brief Title: Heparin and Protamine Titration in Cardiac Surgery Under Minimal Invasive Extracorporeal Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Anna Gkiouliava, PhD candidate, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 7774/16.07.2019
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Cardiopulmonary Bypass
Keywords: anticoagulation; cardiopulmonary bypass

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Individualized heparin and protamine titration (Active Comparator): The device Hemostasis Management System Plus (Medtronic, Minneapolis, MN) will be used to determine the patients' sensitivity to heparin and its concentration in whole blood. Then, it will automatically calculate the necessary dose for anticoagulation during bypass. The protamine dose to eliminate heparin effect will be calculated from the remaining heparin concentration (0.75mg/100 International Units circulating heparin).
  Interventions: Device: Hemostasis Management System Plus
- Activated Clotting Time guided heparin and protamine dose (Active Comparator): Heparin initial dose will be determined according to the patients' weight to achieve a required Activated Clotting Time (ACT) to initiate cardiopulmonary bypass. Subsequent doses of heparin will be administered according to ACT and protamine dose will be calculated from total heparin dose (0.75mg protamine/100 International Units heparin)
  Interventions: Device: Activated Coagulation Timer System Plus

INTERVENTIONS:
Device: Hemostasis Management System Plus — Hemostasis Management System Plus (Medtronic, Minneapolis, MN) is a point of care device useful in the management of heparinization during bypass. It estimates the individual heparin dose response and calculates heparin concentration (IU/ml) in whole blood.
  Arms: Individualized heparin and protamine titration
Device: Activated Coagulation Timer System Plus — The Activated Coagulation Timer System Plus device calculates the Activated Clotting Time (ACT) in seconds.
  Arms: Activated Clotting Time guided heparin and protamine dose

SUMMARY:
During a cardiac surgery under cardiopulmonary bypass it is essential that an appropriate level of anticoagulation is accomplished. To achieve this, the patient is administered heparin. After completion of the surgery, protamine is given to reverse the anticoagulant action of heparin. In this prospective clinical study the researchers will investigate the impact of the two different methods to calculate the required dosage of heparin and protamine; the individualized calculation computed by the Hemostasis Management System Plus (HMS Plus, Medtronic, Minneapolis, MN) device and the weight based. The investigators hypothesize that the aforementioned methods result in different dosages and will elaborate on their impact on postoperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* elective cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

* known blood disorder
* contraindication to heparin administration

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 134 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Total heparin dose | operation duration
  Heparin dose measured in IU
Total protamine dose | At the end of the cardiopulmonary bypass
  Protamine dose measured in mg

SECONDARY OUTCOMES:
Red Blood Cells transfusion | intraoperatively
  Red Blood Cells transfusion measured in units
Red Blood Cells transfusion | 24 hours after the end of the operation
  Red Blood Cells transfusion measured in units
Fibrinogen concentrate transfusion | intraoperatively
  Fibrinogen concentrate transfusion measured in g
Fibrinogen concentrate transfusion | 24 hours after the end of the operation
  Fibrinogen concentrate transfusion measured in g
Prothrombin Complex Concentrate transfusion | intraoperatively
  Prothrombin Complex Concentrate transfusion measured in IU
Prothrombin Complex Concentrate transfusion | 24 hours after the end of the operation
  Prothrombin Complex Concentrate transfusion measured in IU
Platelets transfusion | intraoperatively
  Platelet transfusion measured in units
Platelets transfusion | 24 hours after the end of the operation
  Platelet transfusion measured in units

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Argiriadou, Dr, Study Chair — Associate Professor
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Gkiouliava A, Argiriadou H, Antonitsis P, Goulas A, Papapostolou E, Sarridou D, Karapanagiotidis GT, Anastasiadis K. Individualized heparin monitoring and management reduces protamine requirements in cardiac surgery on minimal invasive extracorporeal circulation; A prospective randomized study. Perfusion. 2024 Nov;39(8):1595-1604. doi: 10.1177/02676591231204284. Epub 2023 Sep 30. PMID 37776194